CLINICAL TRIAL: NCT03938376
Title: Comparison of Micro-ultrasound Targeted Biopsy to mpMRI of Prostate for Detection of Clinically Significant Prostate Cancer
Brief Title: Micro-Ultrasound/Magnetic Resonance Imaging 001
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 19-5042.0
Record Dates: First submitted 2019-04-03; First posted 2019-05-06 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Diagnoses Disease
Keywords: Prostatic Disease; Diagnostic Imaging; Micro-Ultrasound
MeSH Terms: conditions — Prostatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Potential Prostate Cancer: Biopsy naïve patients with rising Prostate Specific Antigen (PSA) results referred by their Urologist for a standard of care (SOC) biopsy.
  Interventions: Diagnostic Test: Micro-Ultrasound guided biopsy

INTERVENTIONS:
Diagnostic Test: Micro-Ultrasound guided biopsy — High-resolution imaging device

SUMMARY:
Micro-ultrasound is a novel real-time imaging modality which maintains the clinical workflow of conventional ultrasound-guided prostate biopsy, while potentially maintaining a similar ability to detect clinically significant prostate cancer (csPCa) to MRI. This prospective trial aims to compare micro-ultrasound to mpMRI in detection of csPCa in the biopsy naïve.

DETAILED DESCRIPTION:
Evidence from a large randomized clinical trial (clinical trials.gov ID NCT02079025), suggests that micro-ultrasound system is more sensitive than conventional transrectal-ultrasound (TRUS) to detect prostate cancer (PCa). the PRI-MUS (prostate risk identification using micro-ultrasound) scoring system was developed and validated to assess the risk of prostate cancer for targeted biopsy with the micro-ultrasound platform, similar to the PIRADS scoring system for suspicious areas on mpMRI. This project will compare micro-ultrasound imaging modality to the current gold-standard imaging for prostate cancer, mpMRI. By applying both modalities to the same patients, the investigators will provide a direct comparison of their screening abilities in terms of sensitivity, specificity, negative predictive value and positive predictive value. It will build evidence to demonstrate that micro-ultrasound may replace MRI/Fusion biopsy in these patients.This project aims to demonstrate that the micro-ultrasound 1) provides more sensitive initial biopsy, reducing the need for repeated procedures, thus lowering the rate of severe sepsis and the number of cancers found after local or regional progression, and 2) reduces the need for mpMRI following initial biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Men with indication for a prostate biopsy will be offered inclusion in the study. Indications for biopsy include clinical suspicion of prostate cancer due to elevated PSA or abnormal digital rectal exam (DRE)

Exclusion Criteria:

* Patients with history of prostate cancer
* Patients with prior prostate biopsies
* Patients who are unwilling or unable to give informed consent
* Patients with contraindication to MRI (i.e. pacemaker, hip prosthesis, severe claustrophobia, brain aneurysm clip, allergy to MRI contrast agent)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Based on the individual's biology, must have suspicion for prostate cancer based on Prostate Specific Antigen (PSA) results.
Study Population: Patients who are referred to confirm negative or positive for diagnosis of prostate cancer based on SOC biopsy, with superior resolution imaging devices. Referral may be indicated in the setting of increased PSA, abnormal DRE and/or abnormality of other serum or urinary tests specific for prostate cancer, for example PHI (Prostate Health Index) and PCA3. The current golden standard imaging for prostate cancer is mpMRI.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
The proportion of csPCa detected for each modality. | 1.5 years
  Micro-ultrasound targeted biopsy will provide a non-inferior sensitivity to detect clinically significant prostate cancer compared to multiparametric MRI.

SECONDARY OUTCOMES:
The proportion of zones of PCa correctly predicted by each modality in the whole-mount pathology specimen for the subset of men selecting radical prostatectomy for treatment. | 1.5 years
  Micro-ultrasound will correctly predict extent of disease in the subset of biopsy subjects who proceed to radical prostatectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeet Ghai, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghai S, Perlis N, Atallah C, Jokhu S, Corr K, Lajkosz K, Incze PF, Zlotta AR, Jain U, Fleming H, Finelli A, van der Kwast TH, Haider MA. Comparison of Micro-US and Multiparametric MRI for Prostate Cancer Detection in Biopsy-Naive Men. Radiology. 2022 Nov;305(2):390-398. doi: 10.1148/radiol.212163. Epub 2022 Jul 19. PMID 35852425